CLINICAL TRIAL: NCT01883635
Title: Dyadic Exercise Intervention for Cancer Survivors and Caregivers
Brief Title: Exercise Intervention for Cancer Survivors and Caregivers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Charles Kamen, Assistant Research Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46413
Record Dates: First submitted 2013-06-05; First posted 2013-06-21 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual Exercise Intervention (Active Comparator): Survivor-only progressive walking and resistance exercise
  Interventions: Behavioral: Survivor-only progressive walking and resistance exercise
- Dyadic Exercise Intervention (Experimental): Dyadic progressive walking and resistance exercise
  Interventions: Behavioral: Dyadic progressive walking and resistance exercise

INTERVENTIONS:
Behavioral: Survivor-only progressive walking and resistance exercise — Daily, home-based, tailored exercise program delivered over the course of 6 weeks to the survivor only
  Other Names: EXCAP
  Arms: Individual Exercise Intervention
Behavioral: Dyadic progressive walking and resistance exercise — Daily, home-based, tailored exercise program delivered over the course of 6 weeks to the survivor and caregiver as a dyad
  Other Names: EXCAP-PA
  Arms: Dyadic Exercise Intervention

SUMMARY:
The purpose of the study is to see whether exercise can improve the health and well-being of cancer survivors. We also want to know about the health and well being of caregivers.

DETAILED DESCRIPTION:
This was a pilot feasibility study to refine our methodology before a larger Phase II trial.

ELIGIBILITY:
Inclusion Criteria for Cancer Survivors:

* Have a diagnosis of cancer (any cancer type excluding squamous and basal cell skin cancers) and have received surgery, chemotherapy, and/or radiation therapy within the last 1-12 months.
* Have a functional capacity rating of 70 or greater on the Karnofsky Performance Scale or a rating of 1 or 0 on the ECOG scale when assessed by a medical oncologist (or physicians designee) following cancer treatments
* Have a caregiver willing to participate int he study
* Be able to read English
* Be 21 years of age or older
* Give written informed consent

Inclusion Criteria for Caregivers:

* Be nominated by a cancer survivor
* Be able to read English
* Be 21 years of age or older
* Give written informed consent

Exclusion Criteria:

* have physical limitations (e.g. cardiorespiratory, orthopedic) contraindicating participation in a low to moderate intensity home based walking and progressive resistance program, as assessed by their medical oncologist, their primary care physician, and/or the study medical monitor.
* For caregivers, be currently undergoing active treatment for cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kamen, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Both cancer survivors and their caregivers were screened, consented, and randomized to one of two intervention arms (Individual Exercise or Dyadic Exercise). 22 cancer survivor/caregiver dyads were recruited (44 individuals).
Groups:
- Individual Exercise Intervention: Progressive walking and resistance exercise treatment, prescribed solely to cancer survivors (daily walking and resistance prescription for 6 weeks)
  Progressive walking and resistance exercise program
- Dyadic Exercise Intervention: Progressive walking and resistance exercise treatment, prescribed to both cancer survivors and their caregivers (daily walking and resistance prescription for 6 weeks)
  Progressive walking and resistance exercise program
Period: Overall Study
Arm/Group | Individual Exercise Intervention | Dyadic Exercise Intervention
Started | 24 | 20
Completed | 20 | 20
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Exercise Intervention | Dyadic Exercise Intervention | Total
Number analyzed (Participants) | 24 | 20 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 35
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.17 (11.05) | 53.90 (12.59) | 55.12 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 19 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 20 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 20 | 44

OUTCOME MEASURES:

1. Primary Outcome: Psychological Distress
Description: Change in psychological distress in the cancer survivor from baseline to 6 weeks, as measured by the Profile of Moods States (POMS) total score. At each time point (baseline and 6 weeks), this questionnaire had a total score range of 0-200, with lower scores signifying less distress. We subtracted the baseline POMS score from the 6 week POMS score; the change score reported below thus has a range from -200 to 200, with lower scores signifying less distress.
Time Frame: Baseline to post-intervention (6 weeks later)
Population: The Primary Outcome analysis looked only at cancer survivors assigned to the Individual Exercise Intervention (n=22) and the Dyadic Exercise Intervention (n=20).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Exercise Intervention | Dyadic Exercise Intervention
Number analyzed (Participants) | 22 | 20
units on a scale | 2.25 (14.24) | -.65 (9.84)
Statistical Analysis 1: Comparison: Individual Exercise Intervention vs Dyadic Exercise Intervention; Test type: Superiority or Other; p = 0.14, t-test, 2 sided; degrees of freedom=40

2. Secondary Outcome: Immune Biomarkers
Description: We measured improvement in immune biomarkers with IL-6, an inflammatory cytokine assessed in the serum of cancer survivors. Numbers presented below are change scores calculated by subtracting baseline IL-6 from post-intervention IL-6 (6 weeks later); lower numbers indicate less inflammation, hypothesized to be linked with better immune function.
Time Frame: Baseline to post-intervention (6 weeks later)
Population: The Secondary Outcome analysis looked only at cancer survivors assigned to the Individual Exercise Intervention (n=22) and the Dyadic Exercise Intervention (n=20).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Individual Exercise Intervention | Dyadic Exercise Intervention
Number analyzed (Participants) | 22 | 20
ng/mL | 1.17 (1.57) | 1.42 (1.24)
Statistical Analysis 1: Comparison: Individual Exercise Intervention vs Dyadic Exercise Intervention; Test type: Superiority or Other; p = 0.65, t-test, 2 sided; degrees of freedom=40

3. Other Pre Specified Outcome: Provision of Social Support
Description: Change in provision of social support from baseline to 6 weeks as reported by the cancer survivor was measured by the Dyadic Support Questionnaire (DSQ). At each time point (baseline and 6 weeks), this questionnaire had a total score range of 0-45, with higher scores signifying more support. We subtracted the baseline score from the 6 week DSQ score; the change score reported below thus has a range from -45 to 45, with higher scores signifying more support.
Time Frame: Baseline to post-intervention (6 weeks later)
Population: This Additional Outcome analysis looked only at cancer survivors assigned to the Individual Exercise Intervention (n=22) and the Dyadic Exercise Intervention (n=20).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Exercise Intervention | Dyadic Exercise Intervention
Number analyzed (Participants) | 22 | 20
units on a scale | -2.90 (1.03) | -1.90 (1.10)
Statistical Analysis 1: Comparison: Individual Exercise Intervention vs Dyadic Exercise Intervention; Test type: Superiority or Other; p = 0.51, t-test, 2 sided; degrees of freedom=40

ADVERSE EVENTS:
Time Frame: 2 years, 3 months
Groups:
- Individual Exercise Intervention - Cancer Survivors; Individual Exercise Intervention - Caregivers: Progressive walking and resistance exercise treatment, prescribed solely to cancer survivors (daily walking and resistance prescription for 6 weeks)
- Dyadic Exercise Intervention - Cancer Survivors; Dyadic Exercise Intervention - Caregivers: Progressive walking and resistance exercise treatment, prescribed to both cancer survivors and their caregivers (daily walking and resistance prescription for 6 weeks)
Arm/Group | Individual Exercise Intervention - Cancer Survivors | Dyadic Exercise Intervention - Cancer Survivors | Individual Exercise Intervention - Caregivers | Dyadic Exercise Intervention - Caregivers
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 1/20 | 0/22 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual Exercise Intervention - Cancer Survivors (N=22) | Dyadic Exercise Intervention - Cancer Survivors (N=20) | Individual Exercise Intervention - Caregivers (N=22) | Dyadic Exercise Intervention - Caregivers (N=20)
1 mm segment depression in EKG (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — 1 mm ST segment depression in Lead II at the end of treadmill test, therefore it was immediately terminated. He was not feeling any discomfort or pain, but because of known heart disease, the exercise physiologist thought it would be best.
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — While exercising, exacerbated her back problems. She has since gone to Chiropractor and massage therapist to help ease pain. Was instructed to stop doing any resistance activity. She will no longer be doing any EXCAP exercises.

LIMITATIONS AND CAVEATS:
First, this was a pilot, Phase I trial, and hence had a limited sample size. This study was conducted in a single geographic region. Finally, we analyzed only two time points: baseline and post-intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No